CLINICAL TRIAL: NCT04532307
Title: Isisekelo Sempilo: HIV Prevention Embedded in Sexual Health: A Pilot Trial to Optimize Peer (Thetha Nami) Delivery of HIV Prevention and Care to Adolescents and Young Adults in Rural KwaZulu-Natal.
Brief Title: Isisekelo Sempilo Trial to Optimize Peer (Thetha Nami) Delivery of HIV Prevention to Young People in Rural KwaZulu-Natal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Africa Health Research Institute (Other)
Responsible Party: Principal Investigator, Maryam Shahmanesh, Associate Professor of Clinical Epidemiology, Africa Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: A00004-TBC
Record Dates: First submitted 2020-03-12; First posted 2020-08-31 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: HIV Prevention
Keywords: HIV prevention; Interventions; Peer support; sexual reproductive health
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care SOC (Experimental): Youth friendly services at Isisekelo Sempilo clinics
  Interventions: Behavioral: Standard of Care SOC
- SRH enhanced Isisekelo Sempilo (Experimental): Self-collected vaginal and urine samples for gonorrhea, chlamydia and trichomonas
  Interventions: Behavioral: Standard of Care SOC; Behavioral: SRH enhanced Isisekelo Sempilo
- Peer-support (Thetha-Nami) (Experimental): Peer support and needs assessment from an area-based peer navigator
  Interventions: Behavioral: Standard of Care SOC; Behavioral: Peer-support (Thetha-Nami)
- SOC + SRH + peer-support (Experimental): Combination of all arms
  Interventions: Behavioral: Standard of Care SOC; Behavioral: SRH enhanced Isisekelo Sempilo; Behavioral: Peer-support (Thetha-Nami); Behavioral: SOC + SRH + peer-support

INTERVENTIONS:
Behavioral: Standard of Care SOC — Research assistants refer the consenting participants to Isisekelo Sempilo adolescent and youth friendly services with HIV testing, treatment if positive and PrEP eligibility screening and offer if negative and family planning
Behavioral: SRH enhanced Isisekelo Sempilo — Self-collected vaginal and urine samples are collected at enrolment. Research assistants then provide an Isisekelo Sempilo clinic referral appointment for results, treatment, HIV testing, sexual health, fertility, and family planning counselling, including the personal benefits of ART and Undetectable=Uninfectious among those infected, and PrEP for those eligible and who are negative.
  Arms: SOC + SRH + peer-support; SRH enhanced Isisekelo Sempilo
Behavioral: Peer-support (Thetha-Nami) — The research assistants refer the participant to a Thetha Nami peer-navigator in their community. Peer navigators will assess their health, social and educational needs, provide mentorship, and help them access the services they need. The peer navigator will facilitate attendance, adherence and retention at the Isisekelo Sempilo clinic.
  Arms: Peer-support (Thetha-Nami); SOC + SRH + peer-support
Behavioral: SOC + SRH + peer-support — A combination of interventions 2 and 3, to include both self-collected STI testing, nurse led testing and counseling, and referral to a Thetha Nami peer navigator to encourage clinic attendance and sexual health promotion.
  Arms: SOC + SRH + peer-support

SUMMARY:
Despite advances in efficacious, efficient and safe biomedical tools to reduce HIV transmission and acquisition the HIV epidemic in South Africa(SA) remains an intractable problem, with the lifetime risk of infection approaching 70% for a 15-year-old girl currently living in northern KwaZulu-Natal, the Africa Health Research Institute(AHRI) research setting. This is in part due to the difficulty in engaging adolescents and youth in HIV interventions. We build on formative work to develop and tailor the interventions to young people's needs. Our findings suggested that young people want to focus on sexual and reproductive health(SRH) and value health-promotion from people of their own age and background (peer-support). In a 2016 population-based study of 15-24-year-olds in the study area we found that one in five had a curable Sexually Transmitted Infection(STI) of which three quarters of did not report any symptoms and would not have been cured with current syndromic management. We also found that home-based self-sampling and treatment for STIs was acceptable and desirable to young people. Based on this we developed and conducted a 6-month pilot of the Isisekelo Sempilo adolescent and youth friendly clinics. These are mobile and fixed clinics that are linked to existing primary care services. The clinics deliver nurse-led HIV-testing, prevention and care integrated with SRH. To date n=337 of those referred from the community(~10%) have attended the clinic. In our setting >85% of school-leavers are unemployed; there are high levels of common mental disorders which increase with age (rising to 32% of those aged 20-22). Systematic reviews have found that community-based delivery of HIV care and peers are effective in supporting HIV care, adherence and virologic suppression. However, none of these interventions have been tested for HIV-prevention and in youth. Based on this we developed and piloted Thetha Nami, an area-based peer-navigator intervention promoting psychosocial well-being in addition to HIV-prevention to young people aged 15-29. Over a four-month period 24-pairs of peer navigators approached 5872, 15-29-year-old men and women, of which 5272 (90%) accepted the needs assessment. We aim to use advances in intervention design and evaluation to answer the question, "will these tailored HIV-prevention interventions developed in partnership with young people arrest the HIV epidemic and improve well-being?"

DETAILED DESCRIPTION:
Study design: We will conduct a 2x2 factorial design intervention pilot trial including 1500 men and women aged 16-29-years old and living in the AHRI surveillance area. The study duration will be 18 months. We will randomly offer one of four combinations of interventions in a factorial trial to 1500 consenting men and women aged 16-29-years old and living in our study area.

Study outcomes: (1) a reduction of the proportion of individuals with infectious HIV (i.e. remaining HIV negative or with an undetectable HIV viral load on treatment if positive) and (2) uptake of comprehensive HIV prevention services, including Pre-Exposure Prophylaxis (PrEP) if negative and antiretroviral (ART) if positive. We will also evaluate uptake of contraception, incidence of pregnancy, mental health and quality of life.

Study Population and Recruitment: Research assistants (RAs) will approach 3000 randomly selected 16-29-year old males and females selected from our demographic surveillance area in their homes. From our experience we expect that 2000 will still be eligible, i.e. aged 16-29 and still living in the surveillance area. RAs will provide information about the study to all eligible participants and consent (in the case of 16-17-year-olds assent with parental consent) them to a) be offered an intervention and b) to be followed up at 12 months to measure the outcome. We anticipate that n=1500 [75% (73-77%)] will consent to participate.

Interventions: a) Standard of Care (SOC): RAs refer participants to adolescent and youth friendly services with family planning, HIV testing and ART if positive and PrEP for those eligible and negative (according to the South African national Department of Health guidelines); b) SRH enhanced arm (Isisekelo Sempilo): Self-collected vaginal and urine samples are collected at enrolment. RAs provide clinic appointment for results, treatment and sexual health promotion and services. These promote fertility and family planning; HIV testing, and benefits of ART including Undetectable=Uninfectious amongst positives and PrEP for those eligible and negative; c) Peer-support (Thetha-Nami): RAs refer the participant to a peer navigator in their community. Peer navigators will assess their health, social and educational needs, provide mentorship, and help them access the services they need. The peer navigator will facilitate attendance, adherence and retention at the clinic; or d) SRH + peer-support.

Data Collection: We will measure linkage to clinical services within 60 days of randomisation and adverse events. At 12 months from enrolment RAs will approach all those who consented at baseline to conduct a tablet-based survey on uptake of HIV prevention and care services, uptake of contraception and pregnancy, mental health (using PHQ9), and quality of life. They will collect dry blood spot for HIV ELISA and HIV viral load, and offer point of-care HIV testing, STI testing and treatment. We will conduct a process evaluation to assess service users and providers and the community experience and any social harms. We will establish the cost of delivering the intervention in each arm.

Analysis: With n=1500 we have the power to show an increase in linkage to clinical services from 10% in SOC to 22% with peer-support or SRH only and 38% with peer-support and SRH. We also have the power to detect a reduction in the proportion of 16-29-year olds with a detectable HIV viral load from 7% to 3.5% at 12 months.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Under 16 years and above 30 years of age, unable to consent

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1743 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of adolescent and youth who have transmissible HIV | 12 months from date of recruitment
  Measured as the proportion of participants who consent to participate with a detectable HIV viral load (>400 copies per ml) 12 months after enrolment per arm
Proportion of adolescents and youth who uptake HIV prevention and treatment services | 60 days
  Measured as the proportion of participants who consent who link to clinical services for HIV testing and PrEP/ART counselling within 60 days per arm
Proportion of adolescents and youth who agree to participate in the trial | 12 months
  Measured as proportion of those who are eligible consenting to offer of interventions who accept interventions and 12 month follow-up
Proportion of adolescents and youth from whom the outcome measure of HIV viral load can be ascertained at 12 months follow-up. | 12 months after enrollment
  Measured as the proportion of all those enrolled that provide dry blood spots for the measurement of HIV (i.e. proportion with an HIV viral load >400 copies per ml) in >75% of those who enrolled at baseline irrespective of engagement in any intervention

SECONDARY OUTCOMES:
Proportion of adolescent and youth who are HIV positive that start antiretroviral treatment | 12 months
  Measured as the proportion who are HIV positive who start treatment per arm; time from randomization to HIV test and treatment initiation per arm.
Proportion of adolescent and youth who are HIV negative who start PrEP and remain negative | 12 months
  Measured as the proportion of those who are PrEP eligible (based on the South African PrEP eligibility criteria) who initiate PrEP when tested negative; Proportion who remain on PrEP at the end of follow-up; and proportion of new HIV diagnosis per arm
Proportion of adolescent and youth that have poor sexual health outcome | 12 months
  Measured as the proportion of enrolled who have a new pregnancy and/or Sexually Transmitted Infection per arm
Proportion of adolescents and youth that have a poor mental health outcome | 12 months from enrolment
  Measured as the proportion screening positive for mental health outcome per arm
Proportion of adolescents and youth that are retained in HIV prevention or care | 12 months from enrolment
  Measured as the Proportion attending at least 3 out of 4 followup visits (month 1, 3, 6, 9) and receiving appropriate HIV test per arm
Proportion of adolescents and youth that have transmissible HIV (on treatment analysis) | 12 months from enrolment
  Measured as the proportion of participants who uptake clinical services who have detectable HIV viral load (>400 copies per ml) 12 months after enrolment per arm

OTHER OUTCOMES:
Process evaluation | 18 months
  Process evaluation of the intervention fidelity; description of acceptability of the intervention components (what works for whom and in which context); unexpected adverse events to the individual and community; and what were the sociodemographic patterns of uptake, retention and adherence?
Costings | 18 months
  What is the cost of the comprehensive SRH component? What is the cost of the peer navigator component? What is the incremental cost per additional person starting and retained in UTT and PrEP at 6 months in each of the arms compared to SoC.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shahmanesh, PhD, Principal Investigator — University College London (UCL) and Africa Health Research Institute (AHRI)
Locations (1):
- AHRI, uMkanyakude, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After study completion data will be stored in Africa Health Research Institute (AHRI) Secure and Safe Data Storage facilities. Data are stored in a database. The database server is located in a secure computer room at the AHRI to which access is restricted to only a few IT professionals. The database is part of the AHRI's Local Area Network, which is protected from outside by a firewall. On the database, the data are stored in MS-SQL Server databases, and access to these is heavily restricted using the features of MS-SQL Server's security subsystem. The AHRI premises are completely surrounded by an electric fence and guarded by a professional security company, 24 hours per day seven days per week. The PI and AHRI data guardian will be responsible for overseeing requests for data sharing. (see below).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available once the primary outcome has been analysed and accepted for publication. We will deposit anonymised IPD data relevant to the analysis in an open access repository at the time of publication.
Access Criteria: The PI and AHRI data guardian will be responsible for overseeing requests for data sharing and that the researchers granted access to the data comply with the terms of the data sharing agreement, which will include honouring any commitments about the use of the data that have been made to participants at the time they granted consent. Researchers will be required to acknowledge the source of the data. The terms will also prohibit researchers attempting to identify participants of the study.

REFERENCES:
- [Derived] Shahmanesh M, Chimbindi N, Busang J, Chidumwa G, Mthiyani N, Herbst C, Okesola N, Dreyer J, Zuma T, Luthuli M, Gumede D, Hlongwane S, Mdluli S, Msane S, Smit T, Molina JM, Khoza T, Behuhuma NO, McGrath N, Seeley J, Harling G, Sherr L, Copas A, Baisley K. Effectiveness of integrating HIV prevention within sexual reproductive health services with or without peer support among adolescents and young adults in rural KwaZulu-Natal, South Africa (Isisekelo Sempilo): 2 x 2 factorial, open-label, randomised controlled trial. Lancet HIV. 2024 Jul;11(7):e449-e460. doi: 10.1016/S2352-3018(24)00119-X. PMID 38925731
- [Derived] Chidumwa G, Chimbindi N, Herbst C, Okeselo N, Dreyer J, Zuma T, Smith T, Molina JM, Khoza T, McGrath N, Seeley J, Pillay D, Tanser F, Harling G, Sherr L, Copas A, Baisley K, Shahmanesh M. Isisekelo Sempilo study protocol for the effectiveness of HIV prevention embedded in sexual health with or without peer navigator support (Thetha Nami) to reduce prevalence of transmissible HIV amongst adolescents and young adults in rural KwaZulu-Natal: a 2 x 2 factorial randomised controlled trial. BMC Public Health. 2022 Mar 7;22(1):454. doi: 10.1186/s12889-022-12796-8. PMID 35255859
- [Derived] Shahmanesh M, Okesola N, Chimbindi N, Zuma T, Mdluli S, Mthiyane N, Adeagbo O, Dreyer J, Herbst C, McGrath N, Harling G, Sherr L, Seeley J. Thetha Nami: participatory development of a peer-navigator intervention to deliver biosocial HIV prevention for adolescents and youth in rural South Africa. BMC Public Health. 2021 Jul 13;21(1):1393. doi: 10.1186/s12889-021-11399-z. PMID 34256725

DOCUMENTS (1):
  • Study Protocol (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT04532307/Prot_000.pdf